CLINICAL TRIAL: NCT00078468
Title: A Phase 2 Open-Label Multicenter Study Of The Garft Inhibitor AG2037 In Patients With Metastatic Colorectal Cancer Who Failed Treatment With A 5-Fluorouracil/Leucovorin Regimen.
Brief Title: Study of the GARFT Inhibitor AG2037 in Patients With Metastatic Colorectal Cancer Who Failed Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A4371004; NCT00085592 (obsolete NCT alias)
Record Dates: First submitted 2004-02-27; First posted 2004-03-02 (Estimated); Last update posted 2006-11-09 (Estimated); Status verified 2006-08

CONDITIONS: Colorectal Neoplasms
MeSH Terms: conditions — Colorectal Neoplasms

INTERVENTIONS:
Drug: PELITREXOL/AG-2037

SUMMARY:
To determine the response rate in patients with metastatic colorectal cancer who failed treatment with a 5-Fluorouracil/Leucovorin regimen and up to one other chemotherapeutic regimen (not including adjuvant chemotherapy).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed metastatic adenocarcinoma of the colon or rectum
* Stage IV or recurrent disease
* Measurable disease
* Disease progression or recurrence during or after completion of prior first-line chemotherapy with fluorouracil and leucovorin calcium (5-FU/LV)
* Prior irinotecan or oxaliplatin as part of the 5-FU/LV regimen or as subsequent therapy allowed
* Only 2 prior regimens for metastatic disease allowed
* One additional regimen as adjuvant therapy allowed provided patient remained disease-free for > 6 months after completion of therapy*
* Newer, targeted investigational agents (e.g., cetuximab or bevacizumab) are not

counted as a chemotherapeutic regimen unless used in combination with a cytotoxic regimen NOTE: *If evidence of failure occurred within < 6 months after completion of adjuvant therapy, patients may have received only 1 additional regimen for metastatic disease

* No active brain metastases (requiring treatment or progressing)

Exclusion Criteria:

* History of blood transfusion within 14 days
* Need of concurrent Administration of allopurinol
* History of Radiotherapy or Chemotherapy within 4 weeks
* Any psychological or sociological condition, addidtive disorder or family problems that might preclude compliance with the protocol
* Any unstable or severe intercurrent medical condition that in the opinion of th einvestigator might interfere with achievement of study objectives
* Receipt of an investigational agent within 28 days prior to first day of dosing with AG-2037
* Pregnant or breast feeding
* Previous treatment with GARFT inhibitors
* History of a malignancy (other than colorectal cancer) excpet those treated with curative intent for skin cancer (other than melanoma) or in situ breast or cervical cancer or those treated with curative intent for any other cancer with no evidence of disease for 5 years
* Active brain metastases (requiring treatment or progression)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56
Dates: Start 2003-12; Study Completion 2004-09

PRIMARY OUTCOMES:
To determine the overall objective response rate (complete and partial responses) of AG-2037 in patients with metastatic colorectal cancer who failed treatment with 5FU/LV regimen and up to one other chemotherapeutic regimen.

SECONDARY OUTCOMES:
To estimate time to progression (TTP).
To evaluate the overall survival (1-year) of patients treated with AG-2037.
To assess changes in patient reported outcomes using health-related quality of life questionnaires.
To evaluate the safety of AG-2037.
To evalutate the PK and PD of AG-2037.
To correlate the various genetic markers of MTAP, folate and purine metabolism with clinical response.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (4):
- United States (4):
  - Pfizer Investigational Site, Poway, California
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, New York, New York

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A4371004&StudyName=Study+of+the+GARFT+Inhibitor+AG2037+in+Patients+with+Metastatic+Colorectal+Cancer+who+Failed+Treatment